CLINICAL TRIAL: NCT02982174
Title: Evaluation of the Signal to Noise Ratio at Various Retinal Layers in Spectral Domain Optical Coherence Tomography (SD OCT) Compared to Swept Source Optical Coherence Tomography (SS OCT)
Brief Title: Evaluation of the Signal to Noise Ratio at Various Retinal Layers
Status: Completed | Type: Observational
Sponsor: Topcon Medical Systems, Inc. (Industry)
Responsible Party: Sponsor
Organization: Topcon Corporation (Industry)
Other Study IDs: Topcon-601-2016
Record Dates: First submitted 2016-11-29; First posted 2016-12-05 (Estimated); Last update posted 2022-06-08 (Actual); Status verified 2022-06

CONDITIONS: Healthy Eyes
Keywords: no known ocular pathology

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Normal Eyes: Subjects with no known ocular diseases will be imaged on the 3D OCT-1 Maestro and DRI OCT Triton
  Interventions: Device: 3D OCT-1 Maestro; Device: DRI OCT Triton

INTERVENTIONS:
Device: 3D OCT-1 Maestro — Image acquisition of the posterior surface of the eye
Device: DRI OCT Triton — Image acquisition of the posterior surface of the eye

SUMMARY:
Compare the signal to noise ratio of each device at various retinal layers.

DETAILED DESCRIPTION:
Compare the signal to noise ratio of each device (SD OCT and SS OCT) at various retinal layers from the same group of subjects

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients > 18 years old who have full legal capacity to volunteer on the date the informed consent is signed.
2. Subjects who can follow the instructions by the clinical staff at the clinical site, and can attend examinations on the scheduled examination date.
3. Subjects who agree to participate in the study.

Exclusion Criteria:

1. History of cataract or ocular surgical procedures that render the cornea opaque or otherwise impact its ability to be imaged using the investigational device.
2. Fixation problems which may prevent obtaining good quality images in either eye.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 30 subjects willing to participate in this study.
Sampling Method: Non-Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2016-12 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Signal to noise ratio between SD OCT and SS OCT | 5 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Wei-Chieh Huang, PhD, Principal Investigator — Topcon Medical Systems, Inc.
Locations (1):
- Topcon Medical Systems Inc., Oakland, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No